CLINICAL TRIAL: NCT01590030
Title: Mesial Incision for Laparoscopic Dermoid Cystectomy: a New Safe and Fertility-sparing Technique
Brief Title: Ovarian Mesial Incision: a New Safe and Fertility-sparing Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Fulvio Zullo, Full Professor, University Magna Graecia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mesial Dermoid Incision
Record Dates: First submitted 2012-04-30; First posted 2012-05-02 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Dermoid Ovarian Cysts

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laparoscopic mesial incision (Experimental)
  Interventions: Procedure: Laparoscopic dermoid cystectomy
- Laparoscopic antimesial incision (Active Comparator)
  Interventions: Procedure: Laparoscopic dermoid cystectomy

INTERVENTIONS:
Procedure: Laparoscopic dermoid cystectomy — Laparoscopy will be performed by pneumoperitoneum with CO2. A complete pelvic examination will be performed to exclude malignant disease. Ovarian capsule will be incised by scissors on mesial side in study group and antimesial side in control group. After cleavage plane identification the cyst enucleation will be completed by atraumatic dissection.

SUMMARY:
The purpose of this study is to evaluate safety and efficacy in terms of spillage risk and fertility-sparing of mesial incision for laparoscopic dermoid cystectomy.

ELIGIBILITY:
Inclusion Criteria:

* reproductive age
* pre-operative findings suggestive for benign tumor
* regular menstrual cycles at least six months before surgery

Exclusion Criteria:

* previous pelvic surgery
* known endocrine disease
* estrogen-progestin use before surgery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2004-09; Primary Completion 2009-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Spillage of intracystic content rate | Intraoperative
Operative times | Immediately at the end of the laparoscopy
  Operative times will be assessed when surgeons will end the laparoscopy, specifically when he will end the suture of the last skin scar.
Chemical peritonitis rate | 1 week after surgery
Intraoperative blood loss | The morning after laparoscopy
  The first patient blood sample will be taken the morning of the surgery, at h 8 am. The day after, it will be taken the second blood sample. Intraoperative blood loss wil be calculated by deducting Hb values of the second hemocrome by the first one.

SECONDARY OUTCOMES:
Ovarian reserve | 3 months and 1 year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Fulvio Zullo, MD, PhD, Principal Investigator — University Magna Graecia
Locations (1):
- Chair of Obstetrics and Gynecology, Catanzaro, CZ, Italy

REFERENCES:
- [Derived] Morelli M, Mocciaro R, Venturella R, Imperatore A, Lico D, Zullo F. Mesial side ovarian incision for laparoscopic dermoid cystectomy: a safe and ovarian tissue-preserving technique. Fertil Steril. 2012 Nov;98(5):1336-40.e1. doi: 10.1016/j.fertnstert.2012.07.1112. Epub 2012 Aug 11. PMID 22884658